CLINICAL TRIAL: NCT03208426
Title: Comparison of the Efficacy of 14-day Sequential Therapy and 10-day Bismuth Quadruple Therapy in the Second Line Therapy for Helicobacter Pylori Infection: A Multi-center Randomized Trial
Brief Title: Sequential Versus Quadruple Therapy in the Second-line Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201611053MINA
Record Dates: First submitted 2017-05-21; First posted 2017-07-05 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Efficacy, Self
MeSH Terms: interventions — Esomeprazole; ribosomal protein S14; Amoxicillin; Clarithromycin; Metronidazole; Tetracycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The technicians who performed the UBT test are blind to the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential therapy for 14 days (Experimental): Sequential therapy for 14 days (experimental) D1-D7: (Nexium, esomeprazole 40mg bid + amoxicillin (Brand name: Amoxicillin Capsule) 1000mg bid) for 7 days D8-D14: (Nexium, esomeprazole 40mg bid + Klaricid XL, clarithromycin 500mg bid + Flagyl, metronidazole 500mg bid) for another 7 days
  Interventions: Drug: Esomeprazole (S14); Drug: Amoxicillin (ST14); Drug: Clarithromycin (ST14); Drug: Metronidazole (ST14)
- bismuth quadruple therapy for 10 days (Active Comparator): Bismuth quadruple therapy for 10 days (active comparator) D1-D10: (Nexium, esomeprazole 40mg bid + KCB F.C. TABLETS, dibismuth trioxide 120mg qid + Flagyl, metronidazole 500mg tid + tetracycline (Brand name: Tetracycline Capsule ) 500mg qid) for 10 days
  Interventions: Drug: Esomeprazole (BQ10); Drug: dibismuth trioxide 120mg (BQ10); Drug: Metronidazole (BQ10); Drug: tetracycline (BQ10)

INTERVENTIONS:
Drug: Esomeprazole (S14) — Nexium, esomeprazole 40mg bid, 14 days
  Other Names: Nexium
  Arms: Sequential therapy for 14 days
Drug: Esomeprazole (BQ10) — Nexium, esomeprazole, 40mg bid for 10 days
  Other Names: Nexium (BQ10)
  Arms: bismuth quadruple therapy for 10 days
Drug: Amoxicillin (ST14) — Day 1-7 amoxicillin (Brand name: Amoxicillin Capsule) 1000mg bid for 7 days
  Other Names: amoxicillin capsule
  Arms: Sequential therapy for 14 days
Drug: Clarithromycin (ST14) — Klaricid-XL, clarithromycin, 500mg, bid, for 7 days, (day 8-14)
  Other Names: Klaricid-XL 500mg
  Arms: Sequential therapy for 14 days
Drug: Metronidazole (ST14) — Flagyl, metronidazole, 500mg bid, for 7 days (day 8-14)
  Other Names: Flagyl
  Arms: Sequential therapy for 14 days
Drug: dibismuth trioxide 120mg (BQ10) — KCB F.C. TABLETS, dibismuth trioxide 120mg qid for 10 days
  Other Names: KCB F.C. TABLETS
  Arms: bismuth quadruple therapy for 10 days
Drug: Metronidazole (BQ10) — Flagyl, metronidazole 500mg tid for 10 days
  Other Names: Flagyl
  Arms: bismuth quadruple therapy for 10 days
Drug: tetracycline (BQ10) — Tetracycline (Brand name: Tetracycline Capsule ) 500mg qid for 10 days
  Other Names: Tetracycline Capsule
  Arms: bismuth quadruple therapy for 10 days

SUMMARY:
Objectives: A recent randomized trial showed that 14-day sequential therapy containing high dose proton pump inhibitor was higher than 95% in the first line treatment. However, whether the 14-day sequential therapy is more effective than 10-day bismuth quadruple therapy remains unknown. Therefore, the investigators aimed to compare the eradication rates and long term re-infection rates of sequential therapy for 14 days versus bismuth quadruple therapy for 10 days in the second line treatment.

DETAILED DESCRIPTION:
This will be a multi-center, open labeled, randomized comparative trial Patients: 240 patients with H. pylori infection who failed after first-line therapy will be eligible

Interventions: eligible patients will be randomized into one of the two groups Group (A): sequential therapy for 14 days (S14)

D1-D7: (esomeprazole 40mg bid + amoxicillin 1000mg bid) for 7 days

D8-D14: (esomeprazole 40mg bid + clarithromycin 500mg bid + metronidazole 500mg bid) for another 7 days

Group (B): bismuth quadruple therapy for 10 days (Q10)

D1-D10: (esomeprazole 40mg bid + dibismuth trioxide 120mg qid + metronidazole 500mg tid + tetracycline 500mg qid) for 10 days

Primary End Point: Eradication rate in the second line treatment according to intention to treat (ITT) analysis in the two treatment groups

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infected patients who fail from first line standard triple therapy with clarithromycin, amoxicillin, and a proton pump inhibitor will be eligible in this study.

Exclusion Criteria:

Patients will be excluded from the study if any one of the following criteria was present:

* children and teenagers aged less than 20 years,
* history of gastrectomy,
* gastric malignancy, including adenocarcinoma and lymphoma,
* previous allergic reaction to antibiotics (bismuth, metronidazole, levofloxacin, tetracycline) and PPI (esomeprazole),
* contraindication to treatment drugs,
* pregnant or lactating women,
* severe concurrent disease, or
* Unwilling to accept random assignment of subjects.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
eradication rate in the second-line treatment according to intention to treat (ITT) analysis | 6 weeks
  Urea breath test will be performed at least 6 weeks after the end of eradication therapy. Successful eradication of H. pylori will be defined as a negative 13C-UBT result. A positive 13C-UBT test will be defined as a delta value of 4 units or greater. All subjects will be asked to stop PPI and H2-blocker for at least two weeks before 13C-UBT.

SECONDARY OUTCOMES:
Incidence of adverse effects in the first line therapy in the two treatment groups | 2 weeks
  At enrollment, the patients will be informed of the common side effects from the studied drugs and they will be asked to record these symptoms during treatment. A standardized interview and questionnaire will be used to assess the adverse events
Eradication rates in the second line treatment according to per protocol (PP) analysis | 6 weeks
  Urea breath test will be performed at least 6 weeks after the end of eradication therapy. Patients not follow the protocol will be excluded for PP analysis.
Changes of gut microbiota in the two treatment groups | 2 weeks, 8 weeks, and 1 year
  the stool specimens before, 2weeks after, 8 weeks after, and 1 year after the treatment will be collected for gut microbiota analysis
Re-infection rate one year after eradication therapy | 1 year
  Urea breath test will be performed 1 year after the end of eradication therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, PhD, Study Chair — National Taiwan University Hospital; Yu-Jen Fang, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- Jyh-Ming Liou, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liou JM, Fang YJ, Chen CC, Bair MJ, Chang CY, Lee YC, Chen MJ, Chen CC, Tseng CH, Hsu YC, Lee JY, Yang TH, Luo JC, Chang CC, Chen CY, Chen PY, Shun CT, Hsu WF, Hu WH, Chen YN, Sheu BS, Lin JT, Wu JY, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Concomitant, bismuth quadruple, and 14-day triple therapy in the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2016 Nov 12;388(10058):2355-2365. doi: 10.1016/S0140-6736(16)31409-X. Epub 2016 Oct 18. PMID 27769562
- [Result] Liou JM, Chen CC, Chen MJ, Chen CC, Chang CY, Fang YJ, Lee JY, Hsu SJ, Luo JC, Chang WH, Hsu YC, Tseng CH, Tseng PH, Wang HP, Yang UC, Shun CT, Lin JT, Lee YC, Wu MS; Taiwan Helicobacter Consortium. Sequential versus triple therapy for the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2013 Jan 19;381(9862):205-13. doi: 10.1016/S0140-6736(12)61579-7. Epub 2012 Nov 16. PMID 23158886